CLINICAL TRIAL: NCT02119325
Title: The Effect of a Nutritional Supplement on Post Prandial Glucose and Lipids in an Adult Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 202180; RH01899 (Other: GSK)
Record Dates: First submitted 2014-04-17; First posted 2014-04-21 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-04

CONDITIONS: Impaired Fasting Glucose
Keywords: fibre; overweight; impaired fasting glucose
MeSH Terms: conditions — Overweight | interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Fibre rich Health Food Drink packed as 30g individual sachet, administered as a single serve in 200 mL of luke warm water
  Interventions: Dietary Supplement: 25% fibre
- Placebo (Placebo Comparator): No Fibre Health Food Drink packed as 25g individual sachet, administered as single serve in 200 mL of luke warm water
  Interventions: Dietary Supplement: 0% fibre

INTERVENTIONS:
Dietary Supplement: 25% fibre — Test is a powdered beverage with an active component of 25% of fibre (resistant maltodextrin)
  Arms: Test
Dietary Supplement: 0% fibre — Placebo is an energy matched powdered beverage
  Arms: Placebo

SUMMARY:
The primary aim of this study is to evaluate the effect of a fibre rich health food drink on the post prandial glucose and triglyceride peak in healthy overweight adults with impaired fasting glucose (IFG). The study is randomised, stratified, double blind, two treatments, two period cross over study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy overweight male and female participants
* Age 18-75 years
* BMI ≥25<35 Kg/m2

Exclusion Criteria:

* Pregnancy/breast-feeding
* Allergy/Intolerance
* Anaemic participants: Hb <10g/dL
* Diabetic participants: fasting blood glucose >125 mg/dL
* Serum Aspartate Transaminase, Alkaline Phosphatase and Serum albumin level 3 times the upper limit of normal range
* Participants on other medications (lipid lowering drugs, oral hypoglycemics)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-09; Primary Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Lambda Therapeutic Research Ltd, Ahmedabad, Gujarat, India

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were mainly recruited from the study site database.
Pre-assignment Details: Of the 210 participants screened, 114 participants were not randomised. The reasons for the same were: not meeting study criteria (n=42), lost to follow-up (n=5), and other reasons (n=67).
Groups:
- Sequence 1: Participants were adminisetered with Test followed by Placebo. Test comprised of a fibre rich health food drink packed as 30g individual sachet, administered as a single serve in 200 mL of luke warm water. The active constituent consisted of 25% fibre (resistant maltodextrin). Placebo was a 'No fibre' health food drink packed as 25g individual sachet, administered as single serve in 200 mL of luke warm water.
- Sequence 2: Participants were administered with Placebo followed by Test. Test comprised of a fibre rich health food drink packed as 30g individual sachet, administered as a single serve in 200 mL of luke warm water. The active constituent consisted of 25% fibre (resistant maltodextrin). Placebo was a 'No fibre' health food drink packed as 25g individual sachet, administered as single serve in 200 mL of luke warm water.
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2
Started | 48 | 48
Completed | 48 | 48
Not Completed | 0 | 0
Period: Washout Period 1
Arm/Group | Sequence 1 | Sequence 2
Started | 48 | 48
Completed | 48 | 47
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2
Started | 48 | 47
Completed | 48 | 47
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Participants
Number analyzed (Participants) | 96
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.9 (7.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 96
Impaired fasting glucose (IFG) status [Number; unit: participants]
  IFG | 26
  No IFG | 70

OUTCOME MEASURES:

1. Primary Outcome: Cmax for Glucose in IFG Status Participants
Description: To evaluate the effect of fibre rich health food drink on post prandial peak (Cmax) for glucose in healthy overweight adults with impaired fasting glucose (IFG)
Time Frame: Blood samples will be taken at -35, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150, 180, 210 & 240 minutes
Population: The per protocol (PP) population was the primary population used for analysis. The PP population included all subjects that fulfil the study entry criteria, receive at least one of the study treatments, have enough plasma samples to estimate the efficacy parameters and are without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Test: Fibre rich Health Food Drink packed as 30g individual sachet, administered as a single serve in 200 mL of luke warm water. The active constituent consisted of 25% fibe (resistant maltodextrin).
Arm/Group | Test | Placebo
Number analyzed (Participants) | 26 | 26
mg/dL | 42.76 (24.229) | 47.40 (23.233)
Statistical Analysis 1: Comparison: Test vs Placebo; H0: There was no difference in the post prandial glucose peak for participants with IFG between the test and placebo. The primary parameter was analysed using a mixed effects model with glucose as dependent variable, treatment and period as fixed effects and subject as random effect; Test type: Superiority or Other; p = 0.0487, ANOVA — Statistical significance at the 5% level was required for both co-primary endpoints in order to progress to formal assessment of secondary endpoints; Difference in Adjusted Mean = -4.64, 95% CI 2-sided [-9.26 to -0.03] — Difference is test minus placebo such that a positive difference means the test has higher Cmax

2. Primary Outcome: Cmax for Triglyceride in IFG Status Participants
Description: To evaluate the effect of fibre rich health food drink on post prandial peak (Cmax) for triglyceride in healthy overweight adults with IFG
Time Frame: Blood samples will be taken at -35, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150, 180, 210 & 240 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Test: Fibre rich Health Food Drink packed as 30g individual sachet, administered as a single serve in 200 mL of luke warm water. The active constituent consisted of 25% fibre (resistant maltodextrin).
Arm/Group | Test | Placebo
Number analyzed (Participants) | 26 | 26
mg/dL | 121.07 (46.484) | 127.85 (72.565)
Statistical Analysis 1: Comparison: Test vs Placebo; H0: There was no difference in the post prandial triglyceride peak for participants with IFG between the test and placebo. The primary parameter was analysed using a mixed effects model with triglyceride as dependent variable, treatment and period as fixed effects and subject as random effect; Test type: Superiority or Other; p = 0.6116, ANOVA — [p-value comment as in outcome 1, analysis 1]; Difference in Adjusted Mean = -6.79, 95% CI 2-sided [-34.02 to 20.44] — Difference is test minus placebo such that a positive difference means the test has higher Cmax

3. Secondary Outcome: Cmax for Glucose in Overweight Healthy Participants
Description: To evaluate the effect of fibre rich health food drink on post prandial peak (Cmax) for glucose in healthy overweight adults
Time Frame: Blood samples will be taken at -35, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150, 180, 210 & 240 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Test | Placebo
Number analyzed (Participants) | 95 | 96
mg/dL | 38.98 (17.687) | 43.64 (19.220)

4. Secondary Outcome: AUC for Glucose in Overweight Healthy Participants
Description: To evaluate the effect of fibre rich health food drink on area under the curve (AUC) for glucose in healthy overweight adults
Time Frame: Blood samples will be taken at -35, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150, 180, 210 & 240 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg*min/dL
Arm/Group | Test | Placebo
Number analyzed (Participants) | 95 | 96
mg*min/dL | 27163.93 (2804.549) | 27329.59 (3040.290)

5. Secondary Outcome: Tmax for Glucose in Overweight Healthy Participants
Description: To evaluate the effect of fibre rich health food drink on the time when maximum post prandial concentration is reached (Tmax) of blood glucose in healthy overweight adults
Time Frame: Blood samples will be taken at -35, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150, 180, 210 & 240 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Test | Placebo
Number analyzed (Participants) | 95 | 96
minutes | 25.74 (15.710) | 25.78 (11.972)

6. Secondary Outcome: Cmax for Triglyceride in Overweight Healthy Participants
Description: To evaluate the effect of fibre rich health food drink on post prandial peak (Cmax) for triglyceride in healthy overweight adults
Time Frame: Blood samples will be taken at -35, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150, 180, 210 & 240 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Test | Placebo
Number analyzed (Participants) | 95 | 96
mg/dL | 126.20 (51.959) | 119.84 (56.151)

7. Secondary Outcome: AUC for Triglycerides in Overweight Healthy Participants
Description: To evaluate the effect of fibre rich health food drink on area under the curve (AUC) for triglycerides in healthy overweight adults
Time Frame: Blood samples will be taken at -35, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150, 180, 210 & 240 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg*min/dL
Arm/Group | Test | Placebo
Number analyzed (Participants) | 95 | 96
mg*min/dL | 59829.76 (27022.972) | 60488.97 (29642.057)

8. Secondary Outcome: Tmax for Triglycerides in Overweight Healthy Participants
Description: To evaluate the effect of fibre rich health food drink on Tmax of triglycerides in healthy overweight adults
Time Frame: Blood samples will be taken at -35, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150, 180, 210 & 240 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Test | Placebo
Number analyzed (Participants) | 95 | 96
minutes | 220.32 (37.115) | 218.75 (30.444)

9. Secondary Outcome: Cmax for RLP Cholesterol in IFG Status Participants
Description: To evaluate the effect of fibre rich health food drink on post prandial Remnant Lipoprotein Cholesterol (RLP Cholesterol) peak (Cmax) in healthy overweight adults with IFG
Time Frame: Blood samples will be taken at -35, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150, 180, 210 & 240 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmole/L
Arm/Group | Test | Placebo
Number analyzed (Participants) | 26 | 26
mmole/L | 0.82 (0.780) | 1.30 (1.265)

10. Secondary Outcome: AUC for RLP Cholesterol in IFG Status Participants
Description: To evaluate the effect of fibre rich health food drink on AUC for RLP Cholesterol in healthy overweight adults with IFG
Time Frame: Blood samples will be taken at -35, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150, 180, 210 & 240 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmole*min/L
Arm/Group | Test | Placebo
Number analyzed (Participants) | 26 | 26
mmole*min/L | 1765.27 (237.951) | 1759.01 (230.544)

11. Secondary Outcome: Tmax for RLP Cholesterol in IFG Status Participants
Description: To evaluate the effect of fibre rich health food drink on Tmax for RLP Cholesterol in healthy overweight adults with IFG
Time Frame: Blood samples will be taken at -35, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150, 180, 210 & 240 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Test | Placebo
Number analyzed (Participants) | 26 | 26
minutes | 124.23 (84.068) | 125.00 (77.006)

12. Secondary Outcome: Cmax for RLP Cholesterol in Overweight Healthy Participants
Description: To evaluate the effect of fibre rich health food drink on post prandial RLP Cholesterol peak (Cmax) in healthy overweight adults
Time Frame: Blood samples will be taken at -35, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150, 180, 210 & 240 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmole/L
Arm/Group | Test | Placebo
Number analyzed (Participants) | 95 | 96
mmole/L | 0.97 (1.009) | 1.33 (1.783)

13. Secondary Outcome: AUC for RLP Cholesterol in Overweight Healthy Participants
Description: To evaluate the effect of fibre rich health food drink on AUC for RLP Cholesterol in healthy overweight adults
Time Frame: Blood samples will be taken at -35, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150, 180, 210 & 240 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmole*min/L
Arm/Group | Test | Placebo
Number analyzed (Participants) | 95 | 96
mmole*min/L | 1856.49 (1049.372) | 1845.29 (904.018)

14. Secondary Outcome: Tmax for RLP Cholesterol in Overweight Healthy Participants
Description: To evaluate the effect of fibre rich health food drink on Tmax of RLP Cholesterol in healthy overweight adults
Time Frame: Blood samples will be taken at -35, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150, 180, 210 & 240 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Test | Placebo
Number analyzed (Participants) | 95 | 96
minutes | 116.84 (77.088) | 130.26 (76.507)

15. Secondary Outcome: Cmax for Insulin in IFG Status Participants
Description: To evaluate the effect of fibre rich health food drink on post prandial peak (Cmax) for insulin in healthy overweight adults with IFG
Time Frame: Blood samples will be taken at -35, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150, 180, 210 & 240 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µIU/mL
Arm/Group | Test | Placebo
Number analyzed (Participants) | 26 | 26
µIU/mL | 190.90 (75.471) | 214.90 (84.080)

16. Secondary Outcome: AUC for Insulin in IFG Status Participants
Description: To evaluate the effect of fibre rich health food drink on AUC for insulin in healthy overweight adults with IFG
Time Frame: Blood samples will be taken at -35, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150, 180, 210 & 240 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µIU*min/mL
Arm/Group | Test | Placebo
Number analyzed (Participants) | 26 | 26
µIU*min/mL | 24920.06 (10299.888) | 27066.11 (10666.718)

17. Secondary Outcome: Tmax for Insulin in IFG Status Participants
Description: To evaluate the effect of fibre rich health food drink on Tmax for insulin in healthy overweight adults with IFG
Time Frame: Blood samples will be taken at -35, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150, 180, 210 & 240 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Test | Placebo
Number analyzed (Participants) | 26 | 26
minutes | 38.46 (23.949) | 39.23 (19.115)

18. Secondary Outcome: Cmax for Insulin in Overweight Healthy Participants
Description: To evaluate the effect of fibre rich health food drink on post prandial peak (Cmax) for insulin in healthy overweight adults
Time Frame: Blood samples will be taken at -35, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150, 180, 210 & 240 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µIU/mL
Arm/Group | Test | Placebo
Number analyzed (Participants) | 95 | 96
µIU/mL | 188.84 (87.184) | 213.42 (100.641)

19. Secondary Outcome: AUC for Insulin in Overweight Healthy Participants
Description: To evaluate the effect of fibre rich health food drink on AUC for insulin in healthy overweight adults
Time Frame: Blood samples will be taken at -35, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150, 180, 210 & 240 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µIU*min/mL
Arm/Group | Test | Placebo
Number analyzed (Participants) | 95 | 96
µIU*min/mL | 21963.63 (10310.800) | 25089.69 (13421.113)

20. Secondary Outcome: Tmax for Insulin in Overweight Healthy Participants
Description: To evaluate the effect of fibre rich health food drink on Tmax for insulin in healthy overweight adults
Time Frame: Blood samples will be taken at -35, 10, 20, 30, 40, 50, 60, 75, 90, 105, 120, 150, 180, 210 & 240 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Test | Placebo
Number analyzed (Participants) | 95 | 96
minutes | 35.58 (24.176) | 36.41 (21.048)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the start of the investigational product, and until one day following last administration of the investigational product.
Arm/Group | Test | Placebo
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/96
Other Adverse Events (participants affected / at risk) | 0/96 | 1/96
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test (N=96) | Placebo (N=96)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.